CLINICAL TRIAL: NCT00836576
Title: A Randomized, Two-way Crossover, Single-dose, Open-label Study to Evaluate the Relative Bioavailability of a Test Tablet Formulation of Benazepril HCl (40 mg), Compared to an Equivalent Dose of a Commercially Available Reference Drug Product (Lotensin®, Novartis Pharmaceuticals Corporation) in 40 Fasted, Healthy, Adult Subjects
Brief Title: Benazepril HCl 40 mg Tablets, Fasting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 01002
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — benazepril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Benazepril HCl 40 mg Tablets
- 2 (Active Comparator)
  Interventions: Drug: Lotensin® 40 mg Tablets

INTERVENTIONS:
Drug: Benazepril HCl 40 mg Tablets — 1 x 40 mg, single-dose fasting
  Arms: 1
Drug: Lotensin® 40 mg Tablets — 1 x 40 mg, single-dose fasting
  Arms: 2

SUMMARY:
The objective of this randomized, single-dose, two-way crossover evaluation is to compare the oral bioavailability of a test benazepril HCl formulation (TEVA Pharmaceutical Industries Ltd.) to an equivalent oral dose of the commercially available benazepril HCl (Lotensin®, Novartis Pharmaceuticals Corporation) in a test population of 40 adults under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male and Female; similar proportions of each preferred.
* Age: At least 18 years.
* Subjects must have a minimum weight of at least 110 pounds.
* Qualifying subjects must be in good health and physical condition as determined by medical history, complete physical examination, and laboratory tests, all obtained within four (4) weeks prior to study start. The subject may not have a history of significant past illness expected to affect the investigation. The normal status of subjects will be confirmed by the following procedures:

  1. Laboratory Tests: Hemoglobin, hematocrit, RBC, WBC, differential count, serum electrolytes (Na, K, Cl), fasting blood glucose, BUN, bilirubin, creatinine, AST, ALT, LDH, alkaline phosphatase, and urinalysis. HIV, Hepatitis B, Hepatitis C, and drugs of abuse testing will be done for screening purposes only. Laboratory values which are greater than ± 20% of the normal range will not qualify unless specifically accepted (with comment) by the Principal Investigator. Results of HIC, Hepatitis B, Hepatitis C, and drugs of abuse must be negative or non-reactive for the subject to qualify for the study. Additional drugs of abuse testing will be done at check-in for each period. Tests are to be negative as a requirement for dosing. Female subjects will have a urine pregnancy test done at screening and prior to each study period at check-in.
  2. Electrocardiogram: A 12-lead electrocardiogram will be obtained for all subjects. The original tracings, plus interpretation, will be included in the case report form packet.
* Subjects must read and sign the Consent Form.

Exclusion Criteria:

* Subjects no complying with the above inclusion criteria must be excluded from the study.
* In addition one of the conditions listed below will exclude a subject from the study:

  1. History of treatment for alcoholism, drug abuse, or substance abuse within the past 24 months.
  2. History of malignancy, stroke, diabetes, cardiac, renal or liver disease, or other serious illness.
  3. History of treatment for asthma within the past five (5) years.
  4. History of treatment for any gastrointestinal disorder within the past five (5) years.
  5. History of neutropenia.
  6. History of hyperkalemia.
  7. History of angioedema.
  8. History of impaired renal function.
  9. History of persistent nonproductive cough.
  10. Females who are pregnant or lactating.
  11. History of hypersensitivity to benazepril HCl, or any angiotensin-converting enzyme (ACE) inhibitor.
* Conditions upon screening which might contraindicate or require that caution be used in the administration of benazepril HCl, including:

  1. Sitting systolic blood pressure below 90 mmHg, or diastolic pressure below 50 mmHg.
  2. Heart rate less than 50 beats per minute after a 5-minute rest in a seated position.
* Inability to read and/or sign the consent form.
* Treatment with any other investigational drug during the four (4) weeks prior to enrollment into the study.
* Subjects who have donated blood within four (4) weeks prior to entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-02; Primary Completion 2001-03 (Actual); Study Completion 2001-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax for Benazepril | Blood samples collected over 96 hours
Bioequivalence based on AUC0-inf for Benazepril | Blood samples collected over 96 hour period
Bioequivalence based on AUC0-t for Benazepril | Blood samples collected over 96 hour period

SECONDARY OUTCOMES:
Cmax results for Benazeprilat | Blood samples collected over 96 hour period
AUC0-inf results for Benazeprilat | Blood samples collected over 96 hour period
AUC0-t results for Benazeprilat | Blood samples collected over 96 hour period

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Siler, M.D., Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Gateway Medical Research, Inc., Saint Charles, Missouri, United States